CLINICAL TRIAL: NCT07331974
Title: A Randomized, Double-blind, Placebo-controlled Trial to Access the Efficacy and Safety of Akkermansia Muciniphila AKM Lab-01 in Participents With Overweigh and Obesity
Brief Title: Efficacy and Safety of Akkermansia Muciniphila AKM Lab-01 for Overweight and Obesity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Moon (Guangzhou) Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MN-AKM-102
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Overweight , Obesity
Keywords: Akkermansia Muciniphila; Obesity; Overweight; Probiotics
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): Subjects receive investigational product AKM Lab-01
  Interventions: Drug: AKM Lab-01
- Placebo (Placebo Comparator): Participants receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AKM Lab-01 — A specific dose of AKM Lab-01 will be administered orally once daily for a period of 3 months.
  Arms: Probiotics
Drug: Placebo — Placebo will be administered orally once daily for a period of 3 months.
  Arms: Placebo

SUMMARY:
This study is designed as a preliminary investigation to evaluate the weight-loss efficacy and safety of AKM Lab-01 in an overweight or obese population. It is an interventional, radomized, double-blind, placebo-controlled clinical trial. Participants who meet the eligibility criteria will be randomly assigned to receive AKM Lab-01 or a matching placebo. The intervention will be administered once daily for 3 months. Baseline metrics, along with blood, urine, and stool samples, will be collected from participants, before and after the AKM Lab-01 intervention. The analysis will focus on changes in body weight, blood lipids, blood glucose, and gut metagenomic profiles (from stool samples). Furthermore, metabolomic analysis of blood and stool samples will be conducted to explore the potential machanisms through which AMK Lab-01 influences body weight.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age: 18-60 years old (inclusive); Gender: male or female.
* 2) Body Mass Index (24.0≤BMI≤40.0 kg/m²).
* 3) Has no taken any medications for metabolic control (e.g., for body weight, blood lipids, or blood glucose) within the past month.
* 4) Has been attempting to manage weight primarily through lifestyle interventions (diet and exercise) for at least one month prior to screening.
* 5) Processes adequate communication and cognitive abilities, is expected to be compliant with long-term medication, and has understood the nature, significance, potential benefits, inconveniences, and risks of the study prior to enrollment.
* 6) For participants of childbearing potential (male or female): Must agree to use at least one medically approved form of contraception (e.g., intrauterine device [IUD], oral contraceptives, or condoms) throughout the trial. For female participants of childbearing potential: Must have a negative serum pregnancy test at screening and must be non-lactating.
* 7) Voluntarily agrees to participate by signing the inform consent form and commits to follow the trial treatment plan and visit schedule.

Exclusion Criteria:

* 1) A clear history of neurological or psychiatric disorders (including epilepsy and dementia).
* 2) Hyperlipidemia due to secondary causes, such as nephrotic syndrome, hepatic diseases, hypothyroidism, or renal failure.
* 3) Concurrent severe medical conditions deemed by the investigator to require immediate treatment, such as severe diabetes mellitus, hypertriglyceridemia, or cerebrovascular disease.
* 4) Concurrent severe primary diseases of the liver, kidney, or hematopoietic system; or individuals with mental illness.
* 5) Participants with a family history of genetically inherited metabolic disorders.
* 6) Participants currently taking hepatotropic medications.
* 7) Participants with a history of prior bariatric surgery.
* 8) Presence of poorly controlled or unstable acute/chronic diseases, including but not limited to:

  * Cardiovascular diseases: Unstable angina, myocardial infarction within the past 6 months, symptomatic congestive heart failure (NYHA Class Ⅱ or higher), severe arrhythmia, ect.
  * Uncontrolled active infectious diseases, malignancies, ect.
* 9) Participants with hepatic or renal insufficiency, defined as:

  * Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) > 2.5 × ULN (Upper Limit of Normal);
  * Serum total bilirubin > 2.5 × ULN;
  * Creatinine (Cr) > 1.5 × ULN.
* 10) Urine amylase ≥ 1.5 × ULN, or any other laboratory abnormality deemed by the investigator to be clinically significant and incompatible with study participation.
* 11) History of acute diabetic complications (e.g., diabetic ketoacidosis or hyperosmolar hyperglycemic state) within the past 3 months.
* 12) History of gastrointestinal surgery within the past year, or the presence of severe, active gastrointestinal disease that is not stabilized and may affect drug absorption, distribution, metabolism, or excretion.
* 13) Know hypersensitivity or allergy to any active ingredient or excipient of the investigational product.
* 14) Use of antibiotic therapy or intake of probiotics/prebiotic supplements within 3 month prior to screening.
* 15) Excessive alcohol consumption (defined as > 30 grams per day for men or > 20 gram, sraems) with the past 10 years.
* 16) pregnant or lactating women.
* 17) Any other medical condition that, in the judgement of the investigator, may put the participant at increased or be aggravated by participation in the study. The specific reason for exclusion based on this criterion must be documented.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Changes in BMI | Baseline, Day 30, Day 60, Day 90
  Changes in BMI from baseline will be assessed
Changes in body weight | Baseline, Day 30, Day 60, Day 90
  Changes in body weight from baseline will be assessed.

SECONDARY OUTCOMES:
Changes in TC | Baseline, Day 90
  Changes in serum TC from baseline will be assessed.
Changes in HbA1c | Baseline, Day 30, Day 90
  Changes in HbA1c from baseline will be assessed.
Changes in Uric Acid | Baseline, Day30, Day90
  Changes in Uric Acid from baseline will be assessed.
Changes in Blood Pressure | Baseline, Day 30, Day 60, Day 90
  Changes of systolic and diastolic blood pressure from baseline will be assessed.
Changes in LDL-C | Baseline, Day 90
  Changes in serum LDL-C from baseline will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Huangpu District People Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided